CLINICAL TRIAL: NCT02442596
Title: Abdominal SepsiS Study: Epidemiology of Etiology and Outcome
Acronym: AbSeS
Status: Completed | Type: Observational
Sponsor: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: ABSES
Record Dates: First submitted 2015-05-05; First posted 2015-05-13 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Intra-Abdominal Infections
Keywords: Abdominal sepsis; Sepsis; Septic shock; Epidemiology; Etiology; Microbiology; Abdomen; Intra-abdominal; Infection; Gastrointestinal tract; Perforation; Peritonitis; Pancreas; Biliary tract; Megacolon
MeSH Terms: conditions — Intraabdominal Infections; Sepsis; Shock, Septic; Infections; Peritonitis; Megacolon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- One Group: This is a prospective observational study, aimed at collecting an adequate dataset on a large cohort of patients admitted to a large number of ICUs.

SUMMARY:
The aim of the project is to perform a multinational, prospective, observational study on IAIs (IntraAbdominal Infections) in critically ill patients; special emphasis will be given to epidemiology and outcomes.

DETAILED DESCRIPTION:
To investigate microbiology and/or drug resistance patterns related to: Geographical region, Source of IAI, Upper GI tract perforation (stomach & duodenum), Lower GI tract perforation (jejunum, ileum, colon, rectum), Primary peritonitis, Peritoneal dialysis-related peritonitis, Intra-abdominal abscess, Pancreatic infection, Biliary tract infection, Typhlitis, Toxic megacolon.

To check the Origin of IAI: community-acquired, early-onset healthcare-associated, late-onset healthcare-associated.

To describe physician's antimicrobial prescription patterns related to a classification grid that stratifies IAIs according to disease expression, community or healthcare origin, and anatomical disruption.

To investigate outcomes (clinical response, need for surgical revision, length of hospitalization, and mortality) related to: Classification of IAI, Severity of acute illness at time of diagnosis (SOFA score) and clinical response after 48-72 hrs. (SOFA score), Processes of care (Time to 1st antimicrobial dose, Time to source control, Type of source control intervention (laparotomy, percutaneous drainage, high volume peritoneal lavage, restoration of anatomy and function), Need for (unplanned) surgical revision (uncontrolled infection source), Frequency of microbiological sampling and delay of results)), Pathogens involved and empirical antimicrobial coverage; special emphasis will be given, to coverage of multidrug resistant Enterobacteriaceae, Pseudomonas aeruginosa, enterococci and Candida species, Duration of antimicrobial therapy, Underlying conditions

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 yrs. of age)
* IAI treated with percutaneous or surgical procedure
* ICU admission (the patient should either be admitted to the ICU because of abdominal sepsis or should be admitted in the ICU for other reasons and subsequently developed abdominal sepsis as a complication during the ICU course)
* Informed consent (if required by local ethics committee)

Exclusion Criteria:

<18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive, adult ICU patients diagnosed with IAI- intra-abdominal infection (either as a primary diagnosis or as a complication during the ICU course) during a 6 months period and with a maximum of 15 cases per unit.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-02 (Actual)

PRIMARY OUTCOMES:
Clinical response | Clinical response at 3 days
Clinical response | Clinical response at 7 days

SECONDARY OUTCOMES:
Surgical revision | within the first week
  For the abdominal sepsis cases that were managed with a surgical intervention (most of them), the need for a surgical revision (re-intervention) within the first week after the initial procedure is considered "failure of initial source control". The need for an additional surgical intervention within the first week will be assessed.
Length of hospitalization | up to 6 months
  Length of ICU stay
Mortality | During the 6 month study period
  Survival status at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Stijn BLOT, Principal Investigator — University Hospital Ghent, Dept. of Internal Medicine; Dirk VOGELAERS, Principal Investigator — University Hospital Ghent, Dept. of Internal Medicine
Locations (1):
- All Centres From All Over the World Willing to Contribute Are Welcome, Brussels, Belgium

REFERENCES:
- [Background] Marshall JC. Intra-abdominal infections. Microbes Infect. 2004 Sep;6(11):1015-25. doi: 10.1016/j.micinf.2004.05.017. PMID 15345234
- [Background] De Waele JJ. Early source control in sepsis. Langenbecks Arch Surg. 2010 Jun;395(5):489-94. doi: 10.1007/s00423-010-0650-1. Epub 2010 Jun 2. PMID 20517699
- [Background] Schein M, Marshall J. Source control for surgical infections. World J Surg. 2004 Jul;28(7):638-45. doi: 10.1007/s00268-004-7505-2. Epub 2004 Jun 8. PMID 15185005
- [Background] Blot S, De Waele JJ. Critical issues in the clinical management of complicated intra-abdominal infections. Drugs. 2005;65(12):1611-20. doi: 10.2165/00003495-200565120-00002. PMID 16060697
- [Background] Rex JH. Candida in the peritoneum: passenger or pathogen? Crit Care Med. 2006 Mar;34(3):902-3. doi: 10.1097/01.CCM.0000202129.19154.64. No abstract available. PMID 16505676
- [Background] de Ruiter J, Weel J, Manusama E, Kingma WP, van der Voort PH. The epidemiology of intra-abdominal flora in critically ill patients with secondary and tertiary abdominal sepsis. Infection. 2009 Dec;37(6):522-7. doi: 10.1007/s15010-009-8249-6. PMID 19669089
- [Background] Swenson BR, Metzger R, Hedrick TL, McElearney ST, Evans HL, Smith RL, Chong TW, Popovsky KA, Pruett TL, Sawyer RG. Choosing antibiotics for intra-abdominal infections: what do we mean by "high risk"? Surg Infect (Larchmt). 2009 Feb;10(1):29-39. doi: 10.1089/sur.2007.041. PMID 19226202
- [Background] Dupont H, Friggeri A, Touzeau J, Airapetian N, Tinturier F, Lobjoie E, Lorne E, Hijazi M, Regimbeau JM, Mahjoub Y. Enterococci increase the morbidity and mortality associated with severe intra-abdominal infections in elderly patients hospitalized in the intensive care unit. J Antimicrob Chemother. 2011 Oct;66(10):2379-85. doi: 10.1093/jac/dkr308. Epub 2011 Jul 25. PMID 21791444
- [Background] Montravers P, Lepape A, Dubreuil L, Gauzit R, Pean Y, Benchimol D, Dupont H. Clinical and microbiological profiles of community-acquired and nosocomial intra-abdominal infections: results of the French prospective, observational EBIIA study. J Antimicrob Chemother. 2009 Apr;63(4):785-94. doi: 10.1093/jac/dkp005. Epub 2009 Feb 5. PMID 19196742
- [Background] Blot S, De Waele JJ, Vogelaers D. Essentials for selecting antimicrobial therapy for intra-abdominal infections. Drugs. 2012 Apr 16;72(6):e17-32. doi: 10.2165/11599800-000000000-00000. PMID 22480338